CLINICAL TRIAL: NCT02534753
Title: A Phase 1, Single-Dose Study to Evaluate the Pharmacokinetics of Intravenous Ascorbic Acid in Healthy Male and Female Volunteers
Brief Title: A Pharmacokinetics Study of Intravenous Ascorbic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGuff Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGP-101
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: Ascor L 500® (Ascorbic Acid Injection, USP)

INTERVENTIONS:
Drug: Ascor L 500® (Ascorbic Acid Injection, USP) — A sterile, solution containing 500 mg ascorbic acid per mL
  Other Names: Ascorbic Acid

SUMMARY:
This is a Phase 1, single-dose study to evaluate the pharmacokinetics of intravenous Ascorbic Acid.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To evaluate the single-dose pharmacokinetics of AA administered intravenously (IV).
2. To evaluate the safety and tolerability of AA administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 18 and 45 years, inclusive.
* Has a body mass index (BMI) between 18 and 32 kg/m2.
* Of sound health and has the ability to understand the requirements of the study and is willing to comply with all study requirements and procedures.

Exclusion Criteria:

* Participates in activities that would not allow accurate evaluation of the pharmacokinetics of Ascorbic Acid
* Medical or physical conditions that would not allow safe participation and/or accurate evaluation of the pharmacokinetics of Ascorbic Acid
* Has participated in an investigational drug study within the 30 days prior to CRU admission.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Concentration of Ascorbic Acid (µM) in plasma | 1 day

SECONDARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) grouped by body system | 1 day
Changes from Baseline in clinical laboratory and vital signs to discharge | 1 day
Changes from pre-dose physical exam findings to discharge | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Damon P Jones, BS/MBA, Study Director — McGuff Pharmaceuticals, Inc.
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States